CLINICAL TRIAL: NCT03365973
Title: A Pilot Study of Pathological Fracture Progression and Related Risk Factors for Patients With Potentially Unstable Spinal Metastases of Breast Cancer
Brief Title: Pathological Fracture in Potentially Unstable Spinal Metastases of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Yuhui Shen, Principal Investigator, Ruijin Hospital
Other Study IDs: RJ2017NO173
Record Dates: First submitted 2017-11-26; First posted 2017-12-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Spinal Metastases; Breast Cancer
Keywords: Pathological Fracture; Indeterminate Instability; Spinal Metastases; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Fractures, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal metastases of breast cancer: Patients with potentially unstable spinal metastases of breast cancer

SUMMARY:
The purpose of this study is to identify potential risk factors for and determine the rate of pathological fracture for patients which having spine metastases from breast cancer and be defined as potentially unstable (SINS 7-12) according to the Spinal Instability Neoplastic Score (SINS). The investigators' analysis will provide robust data about the development of spinal instability and help identify the optimal timing of local surgery treatment.

DETAILED DESCRIPTION:
Considering the concept of spinal instability remains important in the clinical decision-making process for patients with spine metastases, the Spine Oncology Study Group (SOSG) devised an 18-point SINS, which proved reliable and has been widely used in clinical practice. Scores of 0-6, 7-12, 13-18 are considered stable, potentially unstable, and unstable, respectively. Lesions with a low SINS (score 0-6) do not requires surgical interventions, whereas a high SINS (score 13-18) predicts the need for surgical stabilization to restore spinal stability. However, treatment strategy of intermediate SINS (score 7-12) lesions remains ambiguous owing to the uncertainty of spinal stability. With the duration of spinal metastases, some potentially unstable lesions turn to be stable while some turn to be unstable, and several factors such as tumor involvement for vertebral body, radiotherapy may account for different outcomes. Owing to the relatively weaker growth and invasion ability of breast cancer cells compared to other solid tumors such as lung cancer and liver cancer, patients with breast cancer and spinal metastases have longer life expectancy. Reasonable and prompt local surgical intervention to restore spinal stability can achieve pain relief and better quality of life effectively. Moreover, most spinal metastases from breast cancer show lytic or mixed lytic-blastic bone lesions, which exacerbates the spinal stability and results in pathological fracture. Thus, investigators focus on patients which having spinal metastases from breast cancer and an intermediate SINS (score 7-12) to explore the rate of pathological fracture and relevant risk factors. This study will help spine surgeon to identify who could benefit from a prophylactic stabilization procedure with high risk of pathological fracture and when is the best timing of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years, female
* Had a histological confirmation of breast cancer, including all pathological types
* Had a histological or radiological confirmation of spinal metastases from breast cancer
* SINS 7-12

Exclusion Criteria:

* Prior prophylactic stabilization surgery to the spine at current level of interest
* Patients with other malignancies except breast cancer
* Misdiagnosis of spinal metastases from breast cancer confirmed by pathological examination
* Patients without undergoing follow-up on schedule
* Withdraw from the study for any reason

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 120 patients with potentially unstable spinal metastases of breast cancer will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of the pathological fracture of spine | First diagnosis of spinal metastases, every 3 months in the first year after diagnosis, every 6 months after one year after diagnosis. Up to 2 years
  Pathological fracture will be detected using Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Quality of life outcomes measured by EORTC QLQ-C30 questionnaire | First diagnosis of spinal metastases, every 3 months in the first year after diagnosis, every 6 months after one year after diagnosis. Up to 2 years
Quality of life outcomes measured by EORTC QLQ-BM22 questionnaire | First diagnosis of spinal metastases, every 3 months in the first year after diagnosis, every 6 months after one year after diagnosis. Up to 2 years
Pain and functional outcome data measured by Brief Pain Inventory (BPI) questionnaire | First diagnosis of spinal metastases, every 3 months in the first year after diagnosis, every 6 months after one year after diagnosis. Up to 2 years
Spinal stability measured by Spinal Instability Neoplastic Score (SINS) | First diagnosis of spinal metastases, every 3 months in the first year after diagnosis, every 6 months after one year after diagnosis. Up to 2 years
  The Spine Instability Neoplastic Score (SINS) is a comprehensive classification system that can aid in predicting spine stability of neoplastic lesions. The 18-point SINS includes global spinal location of the tumor (score 0-3), type and presence of pain (score 0-3), bone lesion quality (score 0-2), spinal alignment (score 0-4), extent of vertebral body collapse (score 0-3), and posterolateral spinal element involvement (score 0-3). As the SINS increases, the spine stability of neoplastic lesions turns to be worse
Neurologic outcome measured by Frankel grading system | First diagnosis of spinal metastases, every 3 months in the first year after diagnosis, every 6 months after one year after diagnosis. Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuhui Shen, Ph.D., M.D., Principal Investigator — Ruijin Hospital; Weibin Zhang, Ph.D., M.D., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No